CLINICAL TRIAL: NCT05561582
Title: The Effects of Intensity on Exercise-Induced Hypoalgesia During a Knee Extension Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, Abigail Wilson, Assistant Professor, University of Central Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Intensity Exercise (Experimental): Participants will complete a knee extension exercise with weight equivalent to 75% of their 1-repetition maximum for 3 sets of 10 repetitions.
  Interventions: Other: Seated knee extension exercise
- Low Intensity Exercise (Experimental): Participants will complete a knee extension exercise with weight equivalent to 30% of their 1-repetition maximum for 3 sets of 10 repetitions.
  Interventions: Other: Seated knee extension exercise
- Quiet Rest (No Intervention): Participants will sit quietly for two minutes, three times.

INTERVENTIONS:
Other: Seated knee extension exercise — Participants will be seated in a resistance exercise machine. Weight corresponding to the assigned group will be added to the machine. Participants will extend the dominant knee for 3 sets of 10 repetitions.
  Arms: High Intensity Exercise; Low Intensity Exercise

SUMMARY:
The primary purpose of this study is to to compare immediate changes in pressure pain threshold at the exercising muscle (quadriceps) and a non-exercising muscle (upper trapezius) during low and high weight knee extension exercise. Participants will attend one session that consists of pain sensitivity testing, completion of pain-related psychological questionnaires, and random assignment to one of three interventions: 1) knee extension exercise with a high weight, 2) knee extension exercise with a low weight, or 3) quiet rest.

ELIGIBILITY:
Inclusion Criteria:

* Pain-free
* 18-60 years old
* Participant can appropriately perform the knee extension exercise (assessed during screening)

Exclusion Criteria:

* Non-English speaking
* Regular use of prescription pain medications
* Current or history of chronic pain condition
* Currently taking blood-thinning medication
* Systemic medical condition known to affect sensation, such as uncontrolled diabetes or neurological conditions
* Any contraindication to the application of ice, such as: uncontrolled hypertension, cold urticaria, cryoglobulinemia, paroxysmal cold hemoglobinuria, circulatory compromise
* Known presence of cardiovascular, pulmonary, or metabolic disease
* Current use of tobacco products
* Not physically ready to exercise without a medical exam as indicated by the Physical Activity Readiness Questionnaire Plus (PAR-Q+)
* Surgery, injury, or fracture to the lower back or lower extremity within the past 6 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Wilson, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Intensity Exercise | Low Intensity Exercise | Quiet Rest
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Intensity Exercise | Low Intensity Exercise | Quiet Rest | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 60
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.89 (1.74) | 21.50 (2.19) | 21.60 (2.76) | 21.36 (2.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 19 | 49
  Male | 5 | 5 | 1 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 3 | 7
  White | 15 | 17 | 15 | 47
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 60
Pressure Pain Threshold Quadriceps [Mean (Standard Deviation); unit: kilopascals] | 496.16 (175.19) | 499.83 (183.34) | 459.58 (141.85) | 485.19 (169.92)

OUTCOME MEASURES:

1. Primary Outcome: Pressure Pain Threshold
Description: A digital pressure algometer will be applied to the quadriceps and upper trapezius for two trials each. Participants are instructed to say "stop" or "pain" so the stimulus can be terminated "when the sensation first transitions from pressure to pain" (pain threshold). Participants will rate the pain experienced during the threshold testing using a 101-point numeric pain rate scale (NPRS) anchored with 0= no pain to 100= the most intense pain sensation imaginable immediately following each testing time.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: kilopascals
Arm/Group | High Intensity Exercise | Low Intensity Exercise | Quiet Rest
Number analyzed (Participants) | 20 | 20 | 20
kilopascals | 19.11 (77.56) | 48.22 (183.06) | -4.14 (88.66)

2. Secondary Outcome: Conditioned Pain Modulation
Description: Pressure pain threshold after an cold water immersion task will be measured.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: kilopascals
Arm/Group | High Intensity Exercise | Low Intensity Exercise | Quiet Rest
Number analyzed (Participants) | 20 | 20 | 20
kilopascals | -34.44 (98.43) | -21.41 (61.93) | -54.03 (79.56)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | High Intensity Exercise | Low Intensity Exercise | Quiet Rest
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-31): https://cdn.clinicaltrials.gov/large-docs/82/NCT05561582/Prot_SAP_000.pdf